CLINICAL TRIAL: NCT03114527
Title: Phase II Trial of Ribociclib in Combination With Everolimus in Advanced Dedifferentiated Liposarcoma (DDL) and Leiomyosarcoma (LMS)
Brief Title: Phase II Trial of Ribociclib and Everolimus in Advanced Dedifferentiated Liposarcoma (DDL) and Leiomyosarcoma (LMS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAR-096; 17-1013 (Other: Fox Chase Cancer Center Institutional Review Board)
Record Dates: First submitted 2017-03-23; First posted 2017-04-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Soft Tissue Sarcoma
Keywords: Dedifferentiated liposarcoma; DDL; Leiomyosarcoma; LMS; Ribociclib
MeSH Terms: conditions — Sarcoma; Liposarcoma; Leiomyosarcoma | interventions — ribociclib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dedifferentiated Liposarcoma Arm (Experimental): Patients receive ribociclib orally at 300mg/day for 21 days of each 28 day cycle and everolimus 2.5mg orally on a continuous 28 day cycle.
  Interventions: Drug: Ribociclib; Drug: Everolimus
- Leiomyosarcoma Arm (Experimental): Patients receive ribociclib orally at 300mg/day for 21 days of each 28 day cycle and everolimus 2.5mg orally on a continuous 28 day cycle.
  Interventions: Drug: Ribociclib; Drug: Everolimus

INTERVENTIONS:
Drug: Ribociclib — Orally bioavailable, highly selective small molecule inhibitor of CDK4/6
  Other Names: LEE011
Drug: Everolimus — mTOR inhibitor
  Other Names: RAD001; Afinitor

SUMMARY:
This is a two center, 2 arm, Phase II study evaluating the combination of Ribociclib and Everolimus in patients with advanced DDL and LMS who have had at least 1 prior systemic therapy. Patients will be enrolled by sarcoma histology into DDL (Arm A) and LMS (Arm B). The purpose of this study is to determine the anti-tumor activity of this doublet therapy in these patient cohorts. Ribociclib will be administered orally at 300 mg/day 3 weeks on/1 week off. Everolimus will be administered 2.5 mg orally on a continuous 28 day cycle. Clinical and laboratory assessments will be made on day 1, d15 of cycle 1 and 2, and day 1 of each subsequent cycle. Tumor response will be assessed by RECIST 1.1 at (CT or MRI) at week 8, 16, 24 and every 12 weeks thereafter. Study drug administration will continue until disease progression, unacceptable toxicity or withdrawal of consent. Patients will be followed until death or are lost to follow-up for analysis of secondary endpoints.

There will be a 1 step registration process for dedifferentiated liposarcoma patients while patients with leiomyosarcoma will require a 2 step registration process. For step 1 of registration, patients must meet all the eligibility criteria necessary for step 1. For step 2 registration, patients must meet the inclusion criteria necessary for step 2 to be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria Step 1:

* Male or female patients 18 years or older.
* Patients must have locally advanced, metastatic or refractory leiomyosarcoma or dedifferentiated liposarcoma.
* A) Patients enrolled into the dedifferentiated cohort do not require prior systemic therapy (may be naive to systemic therapy). B) Leiomyosarcoma patients must have had at least 1 prior systemic therapy (does not include adjuvant/neoadjuvant therapy in a curative setting). There is no limits on prior number of therapies for either cohort.
* Measurable disease per RECIST 1.1
* Radiological or objective evidence of recurrence or progression on or after the last systemic therapy prior to enrollment.
* Time since the last prior therapy to treat underlying malignancy to start of drug:

  * Cytotoxic chemotherapy: greater than the duration of the most recent cycle of the previous regimen (with a minimum of two weeks for all)
  * Biologic therapy (e.g., antibodies): ≥ four weeks
  * ≥ 5 x t1/2 of a small molecule therapeutic, not otherwise defined above, with a minimum of 2 weeks (including aromatase inhibitors and tamoxifen).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patient has signed the Informed Consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements.
* Patient has adequate bone marrow and organ function as defined by the following laboratory values at screening:

  * Absolute neutrophil count ≥1.5 × 109/L
  * Platelets ≥100 × 109/L
  * Hemoglobin ≥9.0 g/dL
  * Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
  * INR ≤1.5
  * Serum creatinine <1.5 mg/dL or creatinine clearance ≥50 mL/min
  * In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN. If the patient has liver metastases, ALT and AST <5 x ULN
  * Total bilirubin < ULN; or total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome.
  * Fasting plasma glucose <140 mg/dL / 7.7 mmol/L and Glycosylated Hemoglobin (HbA1c) ≤ 8% (both criteria have to be met)
* Fasting serum cholesterol ≤ 300 mg/dl or 7.75 mmol/L and fasting triglycerides ≤ 2.5 × ULN. In case one or both of these thresholds are exceeded, the patient can only be included after initiation of statin therapy and when the above mentioned values have been achieved.
* Must be able to swallow ribociclib and everolimus capsules/tablets.

Exclusion Criteria Step 1:

* Patient has a known hypersensitivity to any of the excipients of Ribociclib or Everolimus.
* Previous treatment with CDK4/6 inhibitors or mTOR inhibitors.
* Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
* Patients with central nervous system (CNS) involvement unless they meet ALL of the following criteria:

  * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
  * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme- inducing anti-epileptic medications for brain metastases.
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patient has a known history of HIV infection (testing not mandatory).
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

  * History of angina pectoris, symptomatic pericarditis, coronary artery bypass graft (CABG) or myocardial infarction within 6 months prior to study entry.
  * Documented cardiomyopathy
  * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
  * History of cardiac failure, significant/symptomatic bradycardia, Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome or any of the following:

    * Known risk to prolong the QT interval or induce Torsade's de Pointes.
    * Uncorrected hypomagnesemia or hypokalemia.
    * Systolic Blood Pressure (SBP) >160 mmHg or <90 mmHg.
    * Bradycardia (heart rate <50 at rest), by ECG or pulse.
    * On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF >450 (based on a mean of 3 ECGs).
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug (see Table 4 for details):

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
  * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
  * Herbal preparations/medications, dietary supplements. Acceptable supplements include multivitamins, vitamin D and calcium
  * Angiotensin-converting enzyme (ACE) inhibitor therapy
* Receipt of a live vaccine within 30 days prior to starting study drug. Examples of live vaccines are: intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid vaccines.
* Patient is currently receiving or has received systemic corticosteroids ≤2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.

  • The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
* Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
* Treatment with an investigational agent within 30 days prior or within 5 half-lives (whichever is longer) before the first dose of the study drug.
* Patient who has received radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to starting study drug, and who has not recovered to Grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥25% of the bone marrow (Ellis, 1961) was irradiated.
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
* Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 4.03 Grade ≤1 (Exception to this criterion: patients with any Grade of alopecia are allowed to enter the study).
* Patient with a Child-Pugh score B or C. See Appendix A.
* Patient has a history of non-compliance to medical regimen or inability to grant consent.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for at least 3 months after completion of treatment. Highly effective contraception methods include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that patient
  * Use of 1 highly effective method of contraception, and 1 additional (barrier) method, at the same time

Highly effective methods: Intra-uterine devices (IUD), Hormonal (birth control pills/oral contraceptives, injectable contraceptives, contraceptive patches, or contraceptive implants) Other effective methods (barrier methods): Latex condom, Diaphragm with spermicide; Cervical cap; Sponge

* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Sexually active males unless they use a condom during intercourse while taking the drug and for 21 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Inclusion Criteria Step 2 (LMS patients only):

- Patients with leiomyosarcoma must have tumors with intact Rb as documented by protein expression by IHC for study entry. Patients without sufficient archival tissue for testing will not be eligible. Please see Section 9.0 for further details on testing and interpretation of results. In the event that a patient has prior sequencing information (i.e. through commercial testing) suggestive of intact Rb, the patient may be included into the study on a case by case basis as determined by the principle investigators. The patient will still be required to submit tissue for Rb determination by IHC, but will not need to wait for these results for study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Antitumor activity of Ribociclib in combination with Everolimus in advanced LMS or DDL | 16 weeks
  Progression free rate

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion
  ORR will be measured by RECIST 1.1.
Progression-free survival (PFS) | Through study completion
  PFS will be measured by RECIST 1.1.
Overall survival (OS) | Through study completion
  OS will be measured from the time of initiation of treatment until death
Number of participants with treatment-related adverse events | Up to 30 days after final treatment on study
  Treatment-related adverse events will be assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, MD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania